CLINICAL TRIAL: NCT05490147
Title: Effect of Low Tidal Volume Ventilation Strategy Combined Goal -Directed Fluid Therapy on Intraoperative Bleeding Undergoing Laparoscopic Major Hepatectomy in Liver Cancer Patients: a Surgeon Blinded Randomized Controlled Study
Brief Title: Effect of Low Tidal Ventilation on Intraoperative Bleeding in Laparoscopic Major Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2206-069-1332
Record Dates: First submitted 2022-07-31; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Ventilator Lung; Liver Cirrhosis; Hepatocellular Carcinoma; Blood Loss, Surgical
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Blood Loss, Surgical | interventions — Tidal Volume; Population Groups

STUDY DESIGN:
Intervention Model Description: a surgeon blinded randomized controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional tidal volume (tidal volume [ml]= ideal body weight [kg]* 10~12) group (Experimental): In the conventional tidal volume group, patients are ventilated with a tidal volume [ml]= ideal body weight [kg]* 10~12 throughout the surgery.
  Interventions: Procedure: conventional tidal volume (tidal volume [ml]= ideal body weight [kg]* 10~12) group
- low tidal (tidal volume [ml]= ideal body weight [kg] * 6~8) volume (Experimental): In the low tidal volume group, patients are ventilated with a tidal volume [ml]= ideal body weight [kg]* 6~8 throughout the surgery.
  Interventions: Procedure: low tidal (tidal volume [ml]= ideal body weight [kg] * 6~8) volume

INTERVENTIONS:
Procedure: conventional tidal volume (tidal volume [ml]= ideal body weight [kg]* 10~12) group — In the conventional tidal volume group, patients are ventilated with a tidal volume [ml]= ideal body weight [kg]* 10~12.
  Arms: conventional tidal volume (tidal volume [ml]= ideal body weight [kg]* 10~12) group
Procedure: low tidal (tidal volume [ml]= ideal body weight [kg] * 6~8) volume — In the low tidal volume group, patients are ventilated with a tidal volume [ml]= ideal body weight [kg]* 6~8.
  Arms: low tidal (tidal volume [ml]= ideal body weight [kg] * 6~8) volume

SUMMARY:
This randomized controlled study's objective is to find a safer mechanical ventilation strategy to reduce intraoperative bleeding in liver cancer patients undergoing laparoscopic major liver resection. The hypothesis is that low tidal volume ventilation in laparoscopic major hepatectomy results in less bleeding.

DETAILED DESCRIPTION:
Patients are randomized into the conventional tidal volume (tidal volume [ml]= ideal body weight [kg]* 10~12) group and low tidal (tidal volume [ml]= ideal body weight [kg] * 6~8) volume group and ventilated accordingly throughout the surgery. All patients undergo general anesthesia with propofol, remifentanil, and rocuronium and are intubated with an endotracheal tube (ID 7.0 for females, ID 7.5 for males). Anesthesia is maintained with sevoflurane, end tidal CO2 is targeted between 30-35mmHg. The radial artery is cannulated and connected to the Flotrac sensor and goal directed fluid therapy is done. The estimated blood loss is checked as the primary outcome. In addition postoperative complications, transfusion amounts, operation time, satisfaction of the surgeon and participants are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma scheduled for laparoscopic major hepatectomy, defined as resection of more than 30% of non-anatomical resection or more than 3 segments

Exclusion Criteria:

* ASA class >4
* patients with chronic obstructive pulmonary disease
* patients with Child-Pugh score C
* patients with arrythmia

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-08-08 (Estimated); Primary Completion 2023-08-08 (Estimated); Study Completion 2023-08-08 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | during surgery
  amount drained from peritoneal cavity - irrigation fluid

SECONDARY OUTCOMES:
postoperative lung complications | op end ~ postoperative 2 weeks
  atelectasis, pneumonia
transfusion amount | op. end ~ postoperative day 3
  RBC, FFP, platelet
postoperative hemoglobin level | op. end ~ postoperative day 3
  postoperative hemoglobin
postoperative total bilirubin level | op. end ~ postoperative day 3
  postoperative total bilirubin level
postoperative PT INR level | op. end ~ postoperative day 3
  postoperative PT INR level
postoperative aspartate aminotransferase level | op. end ~ postoperative day 3
  postoperative aspartate aminotransferase level
postoperative alanine aminotransferase level | op. end ~ postoperative day 3
  postoperative alanine aminotransferase level
postoperative serum creatinine level | op. end ~ postoperative day 3
  postoperative serum creatinine level
operation time | during surgery
  operation time
amount of crystalloids infused | during surgery
  amount of crystalloids infused
Satisfaction scale of the operator and participants | during surgery
  easy 0 - 10 difficult

CONTACTS AND LOCATIONS:
Overall Officials: Seong Mi Yang, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Hendi M, Lv J, Cai XJ. Current status of laparoscopic hepatectomy for the treatment of hepatocellular carcinoma: A systematic literature review. Medicine (Baltimore). 2021 Dec 17;100(50):e27826. doi: 10.1097/MD.0000000000027826. PMID 34918631
- [Background] Nomi T, Fuks D, Govindasamy M, Mal F, Nakajima Y, Gayet B. Risk factors for complications after laparoscopic major hepatectomy. Br J Surg. 2015 Feb;102(3):254-60. doi: 10.1002/bjs.9726. Epub 2014 Dec 17. PMID 25522176
- [Background] Jones RM, Moulton CE, Hardy KJ. Central venous pressure and its effect on blood loss during liver resection. Br J Surg. 1998 Aug;85(8):1058-60. doi: 10.1046/j.1365-2168.1998.00795.x. PMID 9717995
- [Background] Kobayashi S, Honda G, Kurata M, Tadano S, Sakamoto K, Okuda Y, Abe K. An Experimental Study on the Relationship Among Airway Pressure, Pneumoperitoneum Pressure, and Central Venous Pressure in Pure Laparoscopic Hepatectomy. Ann Surg. 2016 Jun;263(6):1159-63. doi: 10.1097/SLA.0000000000001482. PMID 26595124
- [Background] Gao X, Xiong Y, Huang J, Zhang N, Li J, Zheng S, Lu K, Ma D, Yang B, Ning J. The Effect of Mechanical Ventilation With Low Tidal Volume on Blood Loss During Laparoscopic Liver Resection: A Randomized Controlled Trial. Anesth Analg. 2021 Apr 1;132(4):1033-1041. doi: 10.1213/ANE.0000000000005242. PMID 33060490
- [Background] Katz SC, Shia J, Liau KH, Gonen M, Ruo L, Jarnagin WR, Fong Y, D'Angelica MI, Blumgart LH, Dematteo RP. Operative blood loss independently predicts recurrence and survival after resection of hepatocellular carcinoma. Ann Surg. 2009 Apr;249(4):617-23. doi: 10.1097/SLA.0b013e31819ed22f. PMID 19300227
- [Background] Dunki-Jacobs EM, Philips P, Scoggins CR, McMasters KM, Martin RC 2nd. Stroke volume variation in hepatic resection: a replacement for standard central venous pressure monitoring. Ann Surg Oncol. 2014 Feb;21(2):473-8. doi: 10.1245/s10434-013-3323-9. Epub 2013 Oct 23. PMID 24150192
- [Background] Correa-Gallego C, Tan KS, Arslan-Carlon V, Gonen M, Denis SC, Langdon-Embry L, Grant F, Kingham TP, DeMatteo RP, Allen PJ, D'Angelica MI, Jarnagin WR, Fischer M. Goal-Directed Fluid Therapy Using Stroke Volume Variation for Resuscitation after Low Central Venous Pressure-Assisted Liver Resection: A Randomized Clinical Trial. J Am Coll Surg. 2015 Aug;221(2):591-601. doi: 10.1016/j.jamcollsurg.2015.03.050. Epub 2015 Apr 7. PMID 26206652
- [Background] Ratti F, Cipriani F, Reineke R, Catena M, Paganelli M, Comotti L, Beretta L, Aldrighetti L. Intraoperative monitoring of stroke volume variation versus central venous pressure in laparoscopic liver surgery: a randomized prospective comparative trial. HPB (Oxford). 2016 Feb;18(2):136-144. doi: 10.1016/j.hpb.2015.09.005. Epub 2015 Nov 17. PMID 26902132
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Serpa Neto A, Schultz MJ, Gama de Abreu M. Intraoperative ventilation strategies to prevent postoperative pulmonary complications: Systematic review, meta-analysis, and trial sequential analysis. Best Pract Res Clin Anaesthesiol. 2015 Sep;29(3):331-40. doi: 10.1016/j.bpa.2015.09.002. Epub 2015 Sep 18. PMID 26643098